CLINICAL TRIAL: NCT03806647
Title: Taipei Veterans General Hospital
Brief Title: Development and Needs Assessment and Efficiency of Smart Communication System for Patients With ALS (Part 1)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2018-09-001A-1
Record Dates: First submitted 2019-01-14; First posted 2019-01-16 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic lateral sclerosis, ALS, communication, needs
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Communication

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The research is aimed to explore the needs of clinical patients and their caregiver,so as to provide suggestions to the designer of the communication system.

DETAILED DESCRIPTION:
To promote and develop a smart communication system is helpful to patients with amyotrophic lateral sclerosis (ALS),especially for stage 3 and stage 4 (late stage). Through the needs assessment, the research is aimed to explore the needs of clinical patients and their caregiver,so as to provide suggestions to the designer of the communication system.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of ALS
* Taiwanese and used traditional Chinese(Mandarin).
* If they were older than age 20 years.

Exclusion Criteria:

* Frontotemporal dementia, severe depression, or schizophrenia.
* If they cannot complete the questionnaire with researchers or family members help.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with ALS were recruited from ALS clinics(Taipei Veterans General Hospital, Taiwan, R.O.C),20 participants. Participants were eligible for this study if they were diagnosed with definite, probable, probable laboratory-supported, or possible ALS according to the criteria (Brooks et al., 2000).
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-09-01 (Estimated)

PRIMARY OUTCOMES:
Amyotrophic Lateral Sclerosis Supportive Care Needs (ALSSCN) | 2018.10.01~2020.04.31
  The ALSSCN consisted of 37 items with seven domains: physical, psychological, emotional, spiritual, social, informational, and practical needs.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, TW, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided